CLINICAL TRIAL: NCT02245490
Title: BLADDER (BPH, LUTS And Detrusor: Dual Effect Research) Study: A Multicentre, Double-blind, Randomised, Parallel Group, Placebo-controlled Study, Aimed at Characterising the Effect of Tamsulosin on Lower Urinary Tract Symptoms (LUTS) and Detrusor Motor Activity in Patients Affected by Benign Prostatic Hyperplasia (BPH) and Storage Urinary Symptoms
Brief Title: Study to Characterise the Effect of Tamsulosin on Lower Urinary Tract Symptoms (LUTS) and Detrusor Motor Activity in Patients Affected by Benign Prostatic Hyperplasia (BPH) and Storage Urinary Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 527.30
Record Dates: First submitted 2014-09-18; First posted 2014-09-19 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

ARMS (2):
- Tamsulosin (Experimental)
  Interventions: Drug: Tamsulosin HCl controlled release capsules
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo capsule

INTERVENTIONS:
Drug: Tamsulosin HCl controlled release capsules
  Arms: Tamsulosin
Drug: Matching placebo capsule
  Arms: Placebo

SUMMARY:
Study to evaluate the efficacy of tamsulosin on storage symptoms and detrusor motor activity in patients with LUTS suggestive of BPH and relevant storage symptoms

ELIGIBILITY:
Inclusion Criteria:

* Male outpatients aged 50-80 years
* LUTS suggestive of BPH
* Medical history: storage symptoms (frequency, urgency) for at least 6 months
* Urinary Chart:

  * At least 8 micturitions per 24 hours on average, over the week of the screening period (check urinary chart at Visit 2)
  * Urgency (strong desire to void): at least once per 24 hours on average, over the week of the screening period (check urinary chart at Visit 2)
* I-PSS ≥ 13 at randomisation (Visit 3)
* Qmax: > 4 ml/sec at randomisation (Visit 3), with a voiding volume of at least 150 ml
* Prostate Specific Antigen (PSA) < 2.5 ng/ml or between 2.5 and 10 ng/ml, if cancer is ruled out with the usual procedures of each centre (Visit 1; results before Visit 3)
* Written Informed Consent for participation to the study

Exclusion Criteria:

* Patients with a known history or a diagnosis at the time of the screening visit (Visit 1) of the following conditions:
* Urological disturbances

  * Medical history of pelvic surgery
  * Palpable bladder at the physical examination, or residue urinary volume > 400 ml
  * Known neurological bladder disorder
  * Bladder neck stenosis
  * Urethral stricture
  * Bladder or prostatic cancer
  * Bladder stone
  * Severe diverticulum of the bladder
  * Symptomatic urinary tract infection during last month, or recurrent urinary tract infections (more than 2 during last year)
  * Haematuria of unknown origin
  * Diseases which may affect micturition (i.e., diabetes mellitus)
* Cardiovascular diseases (if they occurred in the last 6 months)

  * Myocardial infarction
  * Instable angina
  * Clinically significant ventricular arrhythmias
  * Heart failure (NYHA classes III/IV)
  * Orthostatic hypotension
  * Cerebral stroke
* Neurological diseases (if their severity might compromise the correct performance of the trial)

  * Senile dementia
  * Multiple sclerosis
  * Parkinson's disease
  * Psychiatric disturbances
* Hepatic or renal insufficiency (biochemistry values 15% outside normal lab ranges, being regarded as clinically relevant by the investigator)
* Clinically significant abnormality in the haematological, blood chemistry and urinary values evidenced on the samples taken at the screening visit (Visit 1)
* Patients who are taking or have been taking α-blockers for BPH or for hypertension, or phytotherapy for BPH within the previous 6 weeks
* Patients who were taking or have been taking:

  * α-blockers for BPH or for hypertension within the previous 4 weeks
  * phytotherapy for BPH or mepartricin within the previous 4 weeks
  * finasteride within the previous 6 months
  * anticholinergics within the previous 4 weeks
  * antidiuretics within the previous 4 weeks
  * concomitant drugs which may influence the pharmacodynamic or pharmacokinetic properties of tamsulosin. In particular: α-blockers and mixed α-β-blockers, α- agonists, anti-cholinergics
* Patients who are or have been taking part in a clinical study within the previous 3 months
* Patients who have had hypersensitivity or allergic reactions to previously prescribed α- blocker(s)
* Patients judged by the investigator to be inappropriate for inclusion in the study

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2003-01; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Changes in mean number of micturitions per day | Up to 12 weeks after first drug administration
  As reported in the Urinary Chart

SECONDARY OUTCOMES:
Changes in mean number of urgency episodes per day | Up to 12 weeks after first drug administration
Changes in voided volume per micturition | Up to 12 weeks after first drug administration
Changes in International Prostate Symptom Score (I-PSS) on storage and voiding sub-scores | Up to 12 weeks after first drug administration
Changes in Quality of Life in BPH patients with urinary symptoms (QUIBUS) Italian Score QUIBUS Symptom Score (QUISS) -11 on storage and voiding sub-scores | Up to 12 weeks after first drug administration
Changes in International Index of Erectile Function (IIEF) | Up to 12 weeks after first drug administration
Changes in Uroflowmetry | Up to 12 weeks after first drug administration
Changes in Qmax | Up to 12 weeks after first drug administration
Changes in volume at the first contraction | Up to 12 weeks after first drug administration
Number of unstable contractions | Up to 12 weeks after first drug administration
Maximum amplitude of unstable contractions | Up to 12 weeks after first drug administration
Number of patients with adverse events | Up to 12 weeks after first drug administration